CLINICAL TRIAL: NCT00810459
Title: Trilogy Comparison Study - Pediatrics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philips Respironics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: MR-0713-PTRI-SS
Record Dates: First submitted 2008-12-17; First posted 2008-12-18 (Estimated); Results first posted 2021-02-03 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-01

CONDITIONS: Respiratory Failure
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Trilogy ventilator (Experimental): Trilogy ventilator
  Interventions: Device: Trilogy Ventilator
- Standard of Care (Active Comparator): Participants currently prescribed ventilator
  Interventions: Device: Standard of Care

INTERVENTIONS:
Device: Trilogy Ventilator — Exposure to one hour on the Trilog ventilator
  Arms: Trilogy ventilator
Device: Standard of Care — Exposure of one hour on the Participants prescribed ventilator
  Arms: Standard of Care

SUMMARY:
The objective of this study (Part II) will be to compare the performance of the Trilogy device and a conventional ventilator (participant's current device). Both devices will be set to the participants' current mode and prescription settings.

DETAILED DESCRIPTION:
A. Primary Hypothesis and end-point In patients with respiratory insufficiency, when compared to conventional ventilators, the Trilogy device achieves comparable level of gas exchange (measured as partial pressure of carbon dioxide (CO2) in arterial, venous or capillary blood)and peripheral capillary oxygen saturation, (SpO2) levels during various modes of ventilation.

B. Secondary Hypothesis and end-points In patients with respiratory insufficiency, when compared to conventional ventilators, the Trilogy device achieves comparable breathing pattern (tidal volume, respiratory rate, minute ventilation), hemodynamics (heart rate), and subjective measures of breathing comfort (measured by modified Borg dyspnea scale).

ELIGIBILITY:
Inclusion Criteria:

1. Age > 1years of age; < 18 years of age
2. Greater than 5 kg
3. Considered clinically stable, with low flow oxygen requirements less than 15 LPM (or FIO2 less than 60 %) and PEEP no greater than 10 cm H2O
4. Requiring mechanical ventilation through nasal/facial mask, tracheostomy or endotracheal tube (ET Tube)

Exclusion Criteria:

1. Clinically unstable, i.e.,

   1. Acute Respiratory Failure
   2. Participants with refractory hypotension defined as systolic blood pressure less than 90 mm Hg despite inotropic agents)
   3. Uncontrolled cardiac ischemia or arrhythmias
   4. or as otherwise determined inappropriate for the study as determined by the investigator
2. Patients suffering from metastatic or terminal cancer and patients with do-not-resuscitate orders
3. Pregnancy

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6 (Actual)
Dates: Start 2008-03-10 (Actual); Primary Completion 2009-01-26 (Actual); Study Completion 2009-01-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Mink, MD, Principal Investigator — University of Manitoba
Locations (1):
- University of Manitoba, Winnipeg, Manitoba, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One participant was reconsented to complete the assessment on new software, this participants was not counted twice in the demographics or protocol enrollment.
Groups:
- Trilogy Ventilator First, Then Standard of Care Ventilator: These participants used the Trilogy Ventilator first, then Standard of Care Ventilator
- Standard of Care Ventilator First, Then Trilogy Ventilator: Theses participants used the Standard of Care Ventilator first and then Trilogy Ventilator.
Period: Overall Study
Arm/Group | Trilogy Ventilator First, Then Standard of Care Ventilator | Standard of Care Ventilator First, Then Trilogy Ventilator
Started | 4 | 2
Completed | 4 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants Consented: All participants consented for the study.
Arm/Group | All Participants Consented
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.2 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 5
Region of Enrollment [Number; unit: participants]
  Canada | 6

OUTCOME MEASURES:

1. Primary Outcome: Comparable Level of Gas Exchange (Measured as Partial Pressure of Carbon Dioxide (CO2) in Arterial, Venous or Capillary Blood)
Description: Comparable level of gas exchange (measured as partial pressure of CO2 in arterial, venous or capillary blood)
Time Frame: After one hour of ventilator use
Measure: Mean (Standard Deviation); unit: mEq/L
Groups:
- Trilogy Ventilator: Trilogy ventilator
  Trilogy Ventilator: Exposure to one hour on the Trilogy ventilator
Arm/Group | Trilogy Ventilator | Standard of Care
Number analyzed (Participants) | 6 | 6
mEq/L | 37 (7.5) | 33.3 (11.9)

2. Primary Outcome: Comparable Level of Gas Exchange for Peripheral Capillary Oxygen Saturation (SpO^2)
Description: Comparable level of gas exchange for SpO^2
Time Frame: After one hour of ventilator use
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Trilogy Ventilator | Standard of Care
Number analyzed (Participants) | 6 | 6
mmHg | 94.6 (4.0) | 97.0 (1.9)

3. Secondary Outcome: Heart Rate
Description: heart rate as measured by beats per minute
Time Frame: 60 minutes
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Trilogy Ventilator | Standard of Care
Number analyzed (Participants) | 6 | 6
bpm | 114.5 (26.4) | 103.8 (18.1)

4. Secondary Outcome: Minute Ventilation
Description: Minute ventilation
Time Frame: 60 minutes
Population: One data point not captured
Measure: Mean (Standard Deviation); unit: Lpm
Arm/Group | Trilogy Ventilator | Standard of Care
Number analyzed (Participants) | 5 | 6
Lpm | 4.9 (2.25) | 5.3 (3.2)

5. Secondary Outcome: Tidal Volume
Description: Tidal Volume
Time Frame: 60 minutes
Population: One data point not captured for a participant
Measure: Mean (Standard Deviation); unit: mL/kg
Arm/Group | Trilogy Ventilator | Standard of Care
Number analyzed (Participants) | 5 | 6
mL/kg | 239 (221) | 226 (209)

ADVERSE EVENTS:
Groups:
- Standard of Care Ventilator: Participants currently prescribed ventilator
  Standard of Care: Exposure of one hour on the Participants prescribed ventilator
Arm/Group | Trilogy Ventilator | Standard of Care Ventilator
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No